CLINICAL TRIAL: NCT02536690
Title: The Effect of Remifentanil and Midazolam on Propofol for Loss of Consciousness During Induction of Anesthesia
Brief Title: Remifentanil and Midazolam on Propofol for Loss of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Dr. Koh, Jae Chul, MD, Clinical fellow in department of anesthesiology and pain medicine, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2015-0183-004
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Anesthesia
Keywords: propofol; midazolam; remifentanil; combination; synergic; pharmacodynamics; Loss of consciousness
MeSH Terms: conditions — Unconsciousness | interventions — Propofol; Remifentanil; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group P (Active Comparator): Induction with propofol bolus. Dose will be started at 1 mg/kg and will be adjusted as described in summary.
  Interventions: Drug: Propofol
- Group PR (Active Comparator): Induction with propofol and remifentanil. Remifentanil infusion 0.25 mcg/kg/min for 5 min followed by propofol bolus Propofol dose will be started at 1 mg/kg and will be adjusted as described in summary.
  Interventions: Drug: Propofol; Drug: Remifentanil
- Group PMR (Active Comparator): Induction with propofol, midazolam and remifentanil. Remifentanil infusion 0.25 mcg/kg/min for 5 min followed by midazolam 0.03 mg/kg bolus 1 min after remifentanil infusion start and propofol bolus administration.
  Propofol dose will be started at 1 mg/kg and will be adjusted as described in summary.
  Interventions: Drug: Propofol; Drug: Remifentanil; Drug: Midazolam

INTERVENTIONS:
Drug: Propofol — Propofol bolus dose administration according to the predetermined dose by biased coined design up-and-down study.
  Other Names: Fresofol
Drug: Remifentanil — Remifentanil 0.25 mcg/kg/min infusion for 5 min before propofol administration.
  Other Names: Ultiva
  Arms: Group PMR; Group PR
Drug: Midazolam — Remifentanil 0.25 mcg/kg/min infusion for 5 min before propofol administration followed by midazolam 0.03 mg/kg administration 1 min after remifentanil infusion start.
  Other Names: Vascam
  Arms: Group PMR

SUMMARY:
Propofol in combination with remifentanil or midazolam can result in synergistic or additive effect.

The patients who are scheduled to undergo general anesthesia are enrolled in this study. 120 patients will be randomly allocated to 3 groups(P, PR, PMR). The patients in group P will receive general anesthesia only with propofol and group PR and PMR will receive 0.25 mcg/kg/min remifentanil infusion prior to propofol. The patients in group PMR will receive 0.03 mg/kg bolus dose of midazolam 1 min after start of the remifentanil infusion. 'Success' is defined as loss of both verbal response and eyelash reflex in 2 min after propofol administration. When 'success', the next patient will receive the same dose(in 18/19 probability) or 0.25 mg/kg lower dose(in 1/19 probability) of propofol. When 'failure', the next patient will receive 0.25 mg/kg higher dose of propofol at induction period.

DETAILED DESCRIPTION:
Propofol is a well-known induction agent which can provide sound and quick hypnosis with anti-emetic effects. However, dose dependent hypotension or bradycardia have reported while using this agent. Propofol in combination with remifentanil or midazolam can result in synergistic or additive effect. There are not many studies which provide minimum dose of propofol to induce hypnosis in combination with these agents and advantage of the combination.

The patients who are scheduled to undergo general anesthesia are enrolled in this study. 120 patients will be randomly allocated to 3 groups(P, PR, PMR). Sample size have been decided due to the previous studies which have mentioned 40 participants as a adequate sample size for this biased coin design - up and down study.

After receiving informed consent, patients will be participated in this study. No premedication will be given to the patients before induction. The patients in group P will receive general anesthesia only with propofol and group PR and PMR will receive 0.25 mcg/kg/min remifentanil infusion for 5 min prior to propofol administration. The patients in group PMR will receive 0.03 mg/kg bolus dose of midazolam 1 min after the start of the remifentanil infusion. Initial propofol dose will be 1 mg/kg in each group and the dose will be changed by the result of prior study participant.

'Success' of this study will be defined as loss of both verbal response and eyelash reflex in 2 min after propofol administration. When 'success', the next patient will receive the same dose(in 18/19 probability) or 0.25 mg/kg lower dose(in 1/19 probability) of propofol. When 'failure', the next patient will receive 0.25 mg/kg higher dose of propofol at induction period.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are scheduled to undergo general anesthesia for a surgery.

Exclusion Criteria:

1. ASA class (American Society of Anesthesiologist physical status classification) II or higher
2. Patients with history of allergy or side effects on propofol, remifentanil, midazolam
3. BMI (body mass index) less than 20 or higher than 30
4. Pregnancy
5. Patients taking sedatives or hypnotic agents.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Loss of verbal response and eyelash reflex | 2 minutes after propofol administration
  Checking verbal response by verbal stimulation (yes or no) and reflex by palpation of the levator palpebrae (yes or no).

SECONDARY OUTCOMES:
Mean blood pressure | baseline, propofol administration time (Just after finishing monitoring on the patient in P group, 5 minutes after remifentanil infusion start in PR and PMR group), 1 minute and 2 minutes after propofol administration
  To compare differences among groups in mean blood pressure change (mmHg).
Heart rate | baseline, propofol administration time (Just after finishing monitoring on the patient in P group, 5 minutes after remifentanil infusion start in PR and PMR group), 1 minute and 2 minutes after propofol administration
  To compare differences among groups in heart rate change (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Dong Woo Han, MD, PhD, Study Chair — Department of Anesthesiology and Pain medicine, Gangnam Severance Hospital, Seoul, Korea
Locations (1):
- Gangnam Severance hospital, Seoul, Gangnam-gu, South Korea

REFERENCES:
- [Background] Conway DH, Hasan SK, Simpson ME. Target-controlled propofol requirements at induction of anaesthesia: effect of remifentanil and midazolam. Eur J Anaesthesiol. 2002 Aug;19(8):580-4. doi: 10.1017/s0265021502000935. PMID 12200947
- [Background] Choi SH, Min KT, Lee JR, Choi KW, Han KH, Kim EH, Oh HJ, Lee JH. Determination of EC95 of remifentanil for smooth emergence from propofol anesthesia in patients undergoing transsphenoidal surgery. J Neurosurg Anesthesiol. 2015 Apr;27(2):160-6. doi: 10.1097/ANA.0000000000000094. PMID 25105828
- [Derived] Koh JC, Park J, Kim NY, You AH, Ko SH, Han DW. Effects of remifentanil with or without midazolam pretreatment on the 95% effective dose of propofol for loss of consciousness during induction: A randomized, clinical trial. Medicine (Baltimore). 2017 Dec;96(49):e9164. doi: 10.1097/MD.0000000000009164. PMID 29245361